CLINICAL TRIAL: NCT05229458
Title: Post Marketing Clinical Follow up Study to Evaluate the Performance and Safety of HYALEXO for Pain Relief in Patients Suffering From Osteoarthritis or Degenerative Joint Diseases
Brief Title: Post Marketing Clinical Follow up Study to Evaluate the Performance and Safety of HYALEXO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yooyoung Pharmaceutical Co., Ltd. (Industry)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Other Study IDs: YYDATP-PMCF
Record Dates: First submitted 2022-01-27; First posted 2022-02-08 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Osteoarthritis; Degenerative Joint Disease
MeSH Terms: conditions — Osteoarthritis; Joint Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This trial is a post marketing clinical follow up study, aiming to evaluate the performance and safety of Hyalexo for pain relief in patients suffering from osteoarthritis or degenerative joint diseases.

The study will involve 54 subjects, who will be enrolled in 4 centers in France. The performance outcomes will be evaluated by the koos score, and VAS for pain, while the safety outcomes will be assessed by a safety checklist and by collecting all the adverse events (Adverse Event/Adverse Device Effect/Serious Adverse Event/Serious Adverse Device Effect/Unanticipated Serious Adverse Device Effect/Device Deficiencies) at all visits.

DETAILED DESCRIPTION:
Design:

Open, non-randomised, non-comparative, single group assignment, multicentre study.

Chronogram of visits:

The study foresees the following visits per patient:

* Visit 1 day -3 to day -1: Screening.
* Visit 2 day 0: Baseline visit (1st injection).
* Visit 3 day 7 (± 1 day): Follow up visit and, 2nd injection.
* Visit 4 day 14 (± 2 days): Follow up visit and, 3rd injection.
* Visit 5 day 21 (± 2 days): Follow up visit.
* Visit 6 day 56 (± 2 days): Follow up visit.
* Visit 7 day 98 (± 2 days): Follow up visit.
* Visit 8 day 194 (± 4 days): Final visit.

Patient enrollment and allocation:

After informed consent signature, the patient is considered enrolled. Once the eligibility is established according to inclusion/exclusion criteria the patient will receive a unique patient code and will be allocated to HYALEXO® (the tested medical device). The Investigator must also complete a patient screening log, which reports on all patients who were seen to determine eligibility for inclusion in the study.

Statistical Analysis:

The protocol outlines that a two-sided p-value of 0.05 or less will be used to declare statistical significance for all analyses. Similarly, all confidence intervals will be calculated at the 95% level.

No adjustment for multiplicity will be made to adjust type 1 error rate for secondary endpoints. If necessary, relevant results from other studies already reported in the literature will be considered in the interpretation of results.

The final analysis will be completed after all patients have been exited the study, all queries resolved, and the database have been locked.

If a patient is missing information for one or more variables, the missing data will not be replaced. Quantitative variables (i.e., demographic) if normally distributed will be described through media, standard deviation (SD); variables non-normally distributed will be described using median and range of interquartile.

Considering this clinical trial's design as a longitudinal cohort study, the focus of the performed statistical assessments will be the longitudinal (statistical) analysis.

Primary endpoint, change in Knee injury and Osteoarthritis Outcome Score(KOOS) pain sub-scale score from baseline to 14 weeks visit, will be analysed by performing a Student's t-test for paired data, or a Wilcoxon signed rank test if major deviations from former's test assumptions are recorded. As no missing data imputation on the primary outcome is planned, if such cases arise, a Linear Mixed Model analysis will be performed, to make use of the complete ITT(Intention to treat) population.

Secondary endpoints, all continuous variables in nature, will be assessed by performing ANOVA for repeated measures tests, or ANCOVA for repeated measures tests (if considering covariates like age, sex, BMI, etc.), assuming completeness of data (no missing data). If missingness of data drastically reduces the sample size (e.g., > 5% of patients will be eliminated), a robust statistical analysis method will be employed instead. Such a method, Linear Mixed Models analysis, has the main advantage of making use of the complete ITT population.

The safety analysis will be done on the ITT population.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old(inlcusive≥18years).
* Men or women.
* Patients suffering from painful chronic idiopathic symptomatic degenerative joint diseases(clinical evidence) OR knee osteoarthritis (as defined by the American College of Rheumatology (ACR) criteria); for patients with osteoarthritis at both knees, only the most painful one will be included in the study.
* VAS knee pain≥40mm at screening and 30 days before.
* Patients willing and able to comply with study terms.
* Patients willing to discontinue all other degenerative joint diseases or knee osteoarthritis treatments.

Exclusion Criteria:

* Patients that are unable or unwilling to provide informed consent and/or patients participating in a concurrent clinical trial and/or patients that have participated in a similar clinical trial within the last 30 days.
* Patients with known hypersensitivity to any components of investigational product.
* Patients with infected or severely inflamed joints
* Patients with skin diseases or infections in the area of the injection site.
* Patients with hepatic failure or history thereof.
* Protected persons defined in the following articles of the French Public Health Code:
* L. 1121-5 pregnant women or breastfeeding.
* L. 1121-6: persons deprived of their liberty by a judicial or administrative decision, persons hospitalized without consent and persons admitted to a health or social establishment for purposes other than that of research.
* L. 1121-7: minors.
* L. 1121-8: adults who are subject to legal protection measures or out of state to express their consent.
* L. 1122-1-2: people in emergency situations who cannot give prior consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Four centres in France (about 13 - 14 patients enrolled each; the enrolment is competitive).
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
KOOS for Pain at 12 weeks | 12 weeks
  • Functional assessment of HYALEXO® by KOOS (Knee Injury and Osteoarthritis Outcome score) for Pain subscale at 12 weeks after the last administration of the investigational product, compared to the baseline.
  This was the endpoint used for the sample size calculation.

SECONDARY OUTCOMES:
KOOS for Symptoms, Activity of Daily Living, Sport and Recreation and knee related Quality of life | 1,6,12 weeks and 6 months
  • Functional Assessment of HYALEXO® by KOOS for other Symptoms, Activity of Daily Living (ADL), Sport and Recreation (Sport/Rec) function and knee related Quality of life (QoL) at 1, 6, 12 weeks and 6 months after the last administration of the investigational product, compared to baseline
KOOS for Pain at 1, 6 weeks and 6 months | 1, 6 weeks and 6 months
  • Functional Assessment of HYALEXO® by KOOS for Pain subscale at 1, 6 weeks and 6 months after the last administration of the investigational product, compared to baseline.
Weight-bearing pain using a Visual Analogue Scale(VAS) | 1,6,12 weeks and 6 months
  • Changes in the weight-bearing pain using a Visual Analogue Scale (100 mm - VAS) at 1, 6, 12 weeks and 6 months after the last administration, compared to the baseline.
Changes is rest pain(VAS) | 1,6,12 weeks and 6 months
  • Changes in the rest pain (100 mm - VAS) at 1, 6, 12 weeks and 6 months after the last administration, compared to the baseline.
Changes in motion pain(VAS) | 1,6,12 weeks and 6 months
  • Changes in the motion pain (pain after 15 m walk) (100 mm - VAS) at 1, 6, 12 weeks and 6 months after the last administration, compared to the baseline.
Global Pain Assessment | 1,6,12 weeks and 6 months
  • Patient Global Pain Assessment (100 mm - VAS) at 1, 6, 12 weeks and 6 months after the last administration, compared to the baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Jerome Porterie, Dr, Principal Investigator — Cabinet de Cabinet de Rhumatologie